CLINICAL TRIAL: NCT05318157
Title: Long Term Efficacy of Artemisia Pollen Specific Allergen Immunotherapy in Patients With Seasonal Allergic Rhinitis
Brief Title: Efficacy of Artemisia Pollen Specific Allergen Immunotherapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Tongren Hospital (Other)
Collaborators: Beijing Shijitan Hospital, Capital Medical University (Other); Peking University People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TR-SAR-AIT
Record Dates: First submitted 2022-03-22; First posted 2022-04-08 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-03

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Budesonide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sublingual Immunotherapy group (Experimental)
  Interventions: Drug: AIT drops
- Drugs treatment group (Experimental)
  Interventions: Drug: Clarityne, Rhinocort and Emedastine Difumarate Eye Drops

INTERVENTIONS:
Drug: AIT drops — Once a day
  Arms: Sublingual Immunotherapy group
Drug: Clarityne, Rhinocort and Emedastine Difumarate Eye Drops — The following drugs were permitted as allergy symptoms-relieving medications according to the actual needs in groups: Clarityne, Rhinocort and Emedastine Difumarate Eye Drops, Once a day
  Arms: Drugs treatment group

SUMMARY:
Allergic rhinitis (AR) is a noninfectious inflammatory disease of the nasal mucosa mediated by immunoglobulin E (IgE) after exposure to allergens. Artemisia annua is one of the most important allergen that is responsible for seasonal AR in China during July and October. Allergen specific immunotherapy (AIT) is the only etiological treatment available for AR.

The trial is a randomized, Open label, multicentred trial. A total of 150 subjects with allergic rhinitis caused by Artemisia pollen were recruited and randomized to the immunotherapy group and conversation drugs group.

ELIGIBILITY:
Inclusion Criteria:

* presence of seasonal rhinitis symptoms.
* the TNSS was higher than 6 scores in last autumn pollen season.
* artemisia-specific immunoglobulin E (IgE) levels (ImmunoCAP) at least class 3, and higher than both of ragweed and Humulus IgE levels.
* patients who have been informed of the nature and aims of the study and have given their written consent, willing to comply with the protocol.
* patients who are able to understand the information given and the consent and complete the daily record card.

Exclusion Criteria:

* ulcers, inflammation or trauma in the sublingual part;
* oral diseases / oral allergies;
* had surgery within four weeks before screening evaluation;
* Continuous use of systemic glucocorticoids within four weeks before screening evaluation;
* Any history of severe systemic allergic reaction and eosinophilic esophagitis before screening evaluation;
* Suffering from perennial allergic rhinitis;
* Complicated with chronic rhinitis or sinusitis, nasal polyps;
* In the recent pollen season, rhinitis can be relieved without symptomatic treatment;
* Within 2 years before enrollment, diagnosed with a history of moderate and severe asthma or FEV1 less than 70% of the estimated value;
* Applying β Treatment with receptor blockers (including systemic and local drugs) or angiotensin converting enzyme (ACE) inhibitors;
* Participated in clinical trials of other drugs within one month; Receiving other pollen allergen specific immunotherapy;
* Pregnant and lactating women or those who have pregnancy planning within the past year;
* history of immunosuppressive disease (such as HIV infection history), history of malignancy, history of autoimmune diseases, history of pulmonary tuberculosis, cardiovascular dysfunction, or other serious diseases of other organ systems judged by researchers.
* received pollen allergen specific immunotherapy or are receiving allergen specific immunotherapy within three years.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-10-15 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline symptom scores | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  Symptom change before and after treatment was estimated by Visual analogue scale(VAS) symptom score. The VAS symptom scores ranged from 0 (asymptomatic) to 10 (very severe). Four nasal symptoms (itching, sneezing, rhinorrhoea and nasal obstruction) and two ocular symptoms (ocular itch and watery eyes) were included.
the change of rhinoconjunctivitis quality of life questionnaire (RQLQ) | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  RQLQ score includes 7 aspects and 28 items: nasal symptoms, eye symptoms, non nasal and eye symptoms, behavior problems, sleep, daily activities and emotional reactions. It adopts a 0-6 point design. Among the emotional reactions, 0 point: none at any time; 1 point, not at any time; 2 points, occasionally; 3 points, sometimes; 4 points, often; 5 points, most of the time; 6 points, all the time; In other items: 0 point, not troubled; 1 point, hardly disturbed; 2 points, occasionally troubled; 3 points, moderate distress; 4 points, quite troubled; 5 points, very troubled; 6 points, extremely troubled.

SECONDARY OUTCOMES:
daily medication score | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  medication score in each day during the peak pollen season (ranging from 0 to 3). 0 = no rescue medication uses, 1 = Oral and/or topical non-sedative H1 antihistamines, 2 = Intranasal corticosteroids (Rhinocort) with/without H1 antihistamines, and 3 = Oral corticosteroids with/without intranasal corticosteroids, with/without H1 antihistamines.
combined symptom and medication score, CSMS | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  the daily combined scores of medication and rhinoconjunctivitis symptoms (CSMRS) (ranging from 0 to 6); which was calculated as the combined score of daily average scores of 6 rhinoconjunctivitis symptoms (rhinorrhea, nasal congestion, nasal itching, sneezing, ocular pruritus, and watery eyes) and the daily rescue medication score.
Health economics evaluation | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  Record the treatment cost of patients with allergy related diseases in the period.
adverse events | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  Any adverse event following acupuncture was assessed by physicians and patients. Patients were instructed to record any unexpected signs, symptoms, and feelings during the entire trial period.
The change of biomarkers | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  The levels of neuropeptides; including substance P, vasoactive intestinal peptide (VIP) , neuropeptide Y (NPY)) will be analysed using ELISA. The unit of all these parameters is ng/ml.
The change of cytokine expression | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  Quantitative real-time reverse transcription PCR (qRT-PCR) was used to analyze the mRNA expression levels of the cytokines interleukin-4, interleukin-5, interleukin-13, leukotriene C4, RANTES, tumor necrosis factor-α, thymic stromal lymphopoietin, and EOTAXIN in the nasal mucosa before and after treatment. The qRT-PCR data were processed using the 2-△△CT method.
nasal patency | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  Eccovision acoustic rhinometry was used to measure the nasal cavity volume (NCV) according to standardized recommendations. Measurements of nasal volume were made from the first 2 cm (V2), the first 4 cm (V4), from the first 6 cm (V6), from the segment between 0 and 5 cm (V0-5), and the segment between 0 and 7 cm (V0-7) of the nose. All measurements were performed three times by the same operator, and nasal volumes were calculated as the sum of both nostrils24. In the current study, the change in the nasal cavity volume was measured at 2-5 cm, as this seems to be an important variable for mucosal changes.24 Nasal airway resistance (NAR) was measured by anterior active rhinomanometry in a quiet room at temperature of 25°C and humidity of 70%. NAR was measured at 75 Pa point (R75T).
The change of IgE level | Visit 0: at baseline; Visit 1: at the first year of the high pollen stage; Visit 2: at the second year of the high pollen stage; Visit 3: at ending of 2 years treatment; Visit 4: at the third year of the high pollen stage.
  The levels of sIgE and sIgG will be analysed using Unicap250. The unit of all these parameters is kU/ml.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Beijing Shijitan Hospital, Beijing
  - Beijing TongRen hospitial, Beijing
  - Peking University People's hospital, Beijing